CLINICAL TRIAL: NCT01130337
Title: An Open-label, Multi-center Study to Evaluate the Disease Free Survival Rate of a Perioperative Combination of Capecitabine (Xeloda), Trastuzumab (Herceptin) and Oxaliplatin (XELOX- Trastuzumab) in Patients With Resectable Gastric or Gastro-esophageal Junction Adenocarcinoma
Brief Title: A Study of Capecitabine [Xeloda] in Combination With Trastuzumab [Herceptin] and Oxaliplatine in Patients With Resectable Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25189
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; Trastuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Capecitabine [Xeloda]; Drug: Oxaliplatin; Drug: Trastuzumab [Herceptin]

INTERVENTIONS:
Drug: Capecitabine [Xeloda] — 1.000 mg/m2 orally every 12 hours from day 1 to day 14 of every cycle for 6 cycles
Drug: Oxaliplatin — 130 mg/m2 intravenous infusion day 1 of every cycle
Drug: Trastuzumab [Herceptin] — First dose 8 mg/kg, subsequent cycles 6 mg/kg, intravenously, day of every cycle for 15 cycles

SUMMARY:
This study will evaluate the disease free survival rate of a combination of capecitabine [Xeloda] and oxaliplatin (XELOX) with trastuzumab [Herceptin] in patients with resectable gastric cancer. The combination of Xeloda (orally, 1000 mg/m2 on day 1-14 of every cycle) and Herceptin (intravenously, 8 mg/kg loading dose, then 6 mg/kg on days 1-14 of every cycle) will be administered for three cycles prior to surgery to resect the tumor. If complete resection, R0 or microscopic residual tumor R1 is achieved, patients will continue with three cycles of XELOX and Herceptin and then for completion of 12 months treatment with Herceptin alone. Oxaliplatin will be administered intravenously at a dose of 130 mg/m2 on day 1 in every cycle. The anticipated time on study drug will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Locally advanced resectable HER2-positive gastric or esophagogastric junction adenocarcinoma (Sievert types I, II, III)
* Measurable (RECIST criteria) or assessable disease
* ECOG performance 0-2
* Life expectancy of 12 weeks or more

Exclusion Criteria:

* Immeasurable lesion as the only evidence of disease
* Previous chemotherapy or radiotherapy for gastric neoplasm or some kind of previous surgical resection of the tumor (except diagnostic laparoscopy)
* Concomitant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Spain (22):
  - Elche, Alicante
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Burgos, Burgos
  - Santander, Cantabria
  - Córdoba, Cordoba
  - Granada, Granada
  - Donostia / San Sebastian, Guipuzcoa
  - A Coruña, La Coruña
  - León, Leon
  - Lleida, Lerida
  - Lugo, Lugo
  - Madrid, Madrid
  - Ourense, Orense
  - Vigo, Pontevedra
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Toledo, Toledo
  - Valencia, Valencia
  - Barakaldo, Vizcaya
  - Zaragoza, Zaragoza

REFERENCES:
- [Derived] Rivera F, Izquierdo-Manuel M, Garcia-Alfonso P, Martinez de Castro E, Gallego J, Limon ML, Alsina M, Lopez L, Galan M, Falco E, Manzano JL, Gonzalez E, Munoz-Unceta N, Lopez C, Aranda E, Fernandez E, Jorge M, Jimenez-Fonseca P. Perioperative trastuzumab, capecitabine and oxaliplatin in patients with HER2-positive resectable gastric or gastro-oesophageal junction adenocarcinoma: NEOHX phase II trial. Eur J Cancer. 2021 Mar;145:158-167. doi: 10.1016/j.ejca.2020.12.005. Epub 2021 Jan 20. PMID 33485079

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening period comprised of 35 days. A total of 136 participants were included in the study, of which 36 participants were enrolled and 100 participants discontinued due to screening failures. Abbreviation of AE= adverse event.
Groups:
- Capecitabine+Oxaliplatin+Trastuzumab: Participants received 3 cycles of capecitabine (1,000 milligrams per meter squared [mg/m^2] tablet orally [p.o] twice daily, Days 1-14)/oxaliplatin (130 mg/m^2 as a 120-minute intravenous [IV] infusion, Day 1 of the cycle)/trastuzumab (8 milligrams per kilograms [mg/kg] on Day 1, followed by doses of 6 mg/kg as IV infusion) (XELOX-trastuzumab) as neoadjuvant treatment, every 3 weeks, thereafter, they were assessed for surgery. After surgery, participants received 3 cycles of XELOX-trastuzumab as treatment adjuvant to the surgery, thereafter, another 12 cycles of trastuzumab as monotherapy, was administered every 3 weeks, until disease progression or death.
Period: Overall Study
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Started | 36
Completed | 22
Not Completed | 14
Not completed — Withdrawal by Subject | 3
Not completed — Principal investigator decision | 1
Not completed — Death | 1
Not completed — Disease progression | 1
Not completed — Toxicity, AE/intercurrent disease | 7
Not completed — Surgical resection (R2) | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants.
Groups:
- Capecitabine+Oxaliplatin+Trastuzumab: Participants received 3 cycles of capecitabine (1,000 mg/m^2 tablet p.o twice daily, Days 1-14)/oxaliplatin (130 mg/m^2 as a 120-minute IV infusion Day 1 of the cycle)/trastuzumab (8 mg/kg on Day 1, followed by doses of 6 mg/kg as IV infusion) (XELOX-trastuzumab) as neoadjuvant treatment, every 3 weeks, thereafter, they were assessed for surgery. After surgery, participants received 3 cycles of XELOX-trastuzumab as treatment adjuvant to the surgery, thereafter, another 12 cycles of trastuzumab as monotherapy, was administered every 3 weeks, until disease progression or death.
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.44 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease-free Survival (DFS) at Month 18
Description: DFS was the time elapsed from the time of surgery (for complete resection [R0] participants) until the date on which progression or death from any cause was documented (whichever occured first). Progression was defined as target lesions greater than (>) 20 percent (%) increase in the sum of the longest diameter (SLD) taking as reference the smallest SLD recorded since the treatment started (nadir) and minimum 5 millimeter (mm) increase over the nadir. When the sum becomes very small, increases within the measurement error (2-3 mm) can lead to a 20% increase. Participants who did not present progression and who had not died were censored on the last date on which it was known that there was no progression (last response assessment).
Time Frame: Month 18
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Number analyzed (Participants) | 36
percentage of participants | 76.12 [57.72 to 87.32]

2. Secondary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: pCR was defined as an absence of any invasive cancer cell of the primary tumor after the time of major neoadjuvant chemotherapy, with or without surgery.
Time Frame: Between Days 7 and 21 of the 3rd cycle of neoadjuvant treatment, thereafter, every 9 weeks during adjuvant treatment and then after adjuvant treatment every 3 months until Month 25
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Number analyzed (Participants) | 36
percentage of participants | 8.33 [1.75 to 22.47]

3. Secondary Outcome: Percentage of Participants With Complete Tumor Resection (R0)
Description: R0 resection was defined as having performed a complete resection of the tumor with adequate tumor-free margins and regional lymph node extirpation.
Time Frame: as for outcome 2
Population: ITT population. Here "number of participants analyzed" included those who underwent surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Number analyzed (Participants) | 31
percentage of participants | 90.32 [74.25 to 97.96]

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: An objective response was defined as either a complete response (CR) or a partial response (PR). Using the Response Evaluation Criteria in Solid Tumors (RECIST), CR was defined as the disappearance of all target lesions and all non-target lesions, normalization of tumor marker level, and no new lesions. PR was defined as the disappearance of all target lesions and persistence of greater than or equal to (≥) 1 non-target lesions and/or the maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diameter of target lesions, and no new lesions or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Number analyzed (Participants) | 36
percentage of participants | 38.89

ADVERSE EVENTS:
Time Frame: Before Day 1 of each cycle until Month 25
Description: The safety analysis included all participants in the ITT population who received at least 1 dose of the study drugs.
Arm/Group | Capecitabine+Oxaliplatin+Trastuzumab
Serious Adverse Events (participants affected / at risk) | 22/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine+Oxaliplatin+Trastuzumab (N=36)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Localised intra-abdominal fluid collection (Gastrointestinal disorders) | 2 (2)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine+Oxaliplatin+Trastuzumab (N=36)
Anaemia (Blood and lymphatic system disorders) | 11 (13)
Neutropenia (Blood and lymphatic system disorders) | 7 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (16)
Abdominal pain (Gastrointestinal disorders) | 9 (12)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 29 (68)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 5 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 17 (29)
Vomiting (Gastrointestinal disorders) | 15 (26)
Asthenia (General disorders) | 24 (61)
Mucosal inflammation (General disorders) | 8 (9)
Pyrexia (General disorders) | 10 (13)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Ejection fraction decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 15 (30)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysaesthesia (Nervous system disorders) | 7 (18)
Dysgeusia (Nervous system disorders) | 3 (5)
Neuropathy peripheral (Nervous system disorders) | 6 (9)
Neurotoxicity (Nervous system disorders) | 10 (16)
Paraesthesia (Nervous system disorders) | 6 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.